CLINICAL TRIAL: NCT02288780
Title: Transthoracic Echocardiographic Evaluation of the Cardiac Function During Transurethral Resection of Prostate in Elderly Patients
Status: Terminated | Type: Observational
Why Stopped: It was difficult to proceed with the study according to the protocol, the research was terminated early.
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2014-0734
Record Dates: First submitted 2014-10-30; First posted 2014-11-11 (Estimated); Last update posted 2019-03-18 (Actual); Status verified 2019-03

CONDITIONS: BPH

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Control: BPH patients with normal diastolic function
- Diastolic dysfunction: BPH patients with preoperative diastolic dysfunction

SUMMARY:
Transurethral resection of the prostate (TURP) is a standard surgical treatment for benign prostatic hyperplasia (BPH). Non-conductive irrigation fluid is used to maintain good visibility of the operating field during resection of the prostate. Absorption of this hypotonic solution into the bloodstream can cause fluid overload and dilutional hyponatremia, resulting in adverse cardiovascular and central nervous system effects, transurethral resection (TUR) syndrome. BPH is common in elderly men above 60 years old. These aged people commonly have diastolic impairment by normal physiologic change without consistent symptom. This study aimed to evaluate the cardiac function focused mainly diastolic function during TURP with transthoracic echocardiography. Also, we will focus the effets of amount of irrgation fluid on left ventricular diastolic function in patients with pre-existing diastolic dysfunction.

ELIGIBILITY:
Inclusion Criteria:

1. Above 65years of age
2. American Society of Anesthesiologists (ASA) Physical Status I, II, III.
3. undergoing transurethral resection of the prostate(TURP)"

Exclusion Criteria:

1. severe coagulopathy or bleeding disorder(platelet count<75000, PT INR >1.2)
2. short stature (under 150 cm)
3. underwent coronary artery bypass graft
4. contraindications of regional anesthesia "

Ages: 65 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: BPH patients with/without preoperative diastolic dysfunction
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2015-05-01 (Actual); Study Completion 2015-05-01 (Actual)

PRIMARY OUTCOMES:
diastolic function by TTE | The participants will be followed for the duration of surgery (TURP), an expected average of 1 hour.